## Study Title:

Development and Evaluation of a Mindfulness-Based Emotional Eating Reduction Program (MBEER)

## **NCT Number:**

[To be filled after ClinicalTrials.gov registration]

## **Document Date:**

May 21, 2023

## **Informed Consent Form**

- I declare that I am over the age of 18.
- I acknowledge that the Mindfulness-Based Emotional Eating Reduction Program is not a diet program and is not intended for weight gain, weight loss, or weight management. I understand that I am responsible for my own physiological and psychological health throughout the program.
- I understand that I am enrolling in a training program that includes physical, emotional, and psychological activities, and that such programs may inherently involve risks.
- To the best of my knowledge, I declare that I do not have any physical, emotional, or psychological conditions that would prevent me from participating in this training.
- I understand that during the Mindfulness-Based Emotional Eating Reduction

  Program, personal matters may inevitably arise, but this training is aimed at
  increasing awareness related to eating behaviors and does not adequately address
  personal psychological issues.
- I acknowledge that the training staff cannot continuously monitor my physical, emotional, or psychological condition. Therefore, I accept responsibility for evaluating any risks posed by a particular activity and for choosing behavior that is safe for me.
- I accept responsibility for completing the assignments and tasks given as part of the program's evaluation process.
- I understand that this study, which I voluntarily applied to participate in, is not a form of therapy or psychological support, nor does it provide dietary consultation.

- I acknowledge that participation in at least 6 weeks of the Mindfulness-Based Emotional Eating Reduction Program is mandatory and that otherwise, I will not be eligible to receive a certificate of participation. I understand that the certificate does not grant me any practitioner qualification.
- I acknowledge that at any stage of the program, the program facilitator has the authority to decide whether I may continue participation, should they deem it necessary, and I accept that their decision will be binding.

| Name Surname: |
|---------------|
| Date: |
| Signature: |